CLINICAL TRIAL: NCT02749058
Title: Capsulectomy vs Capsulotomy in Total Hip Arthroplasty. Clinical Outcomes and Proprioception Evaluation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gianfranco Fraschini, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAP_Feb16
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Hip Arthrosis
Keywords: capsulectomy; capsulotomy
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsulectomy (Other): Procedure: Capsulectomy in Direct Anterior Total Hip Arthroplasty
  Interventions: Procedure: Capsulectomy in Direct Anterior Total Hip Arthroplasty
- Capsulotomy (Other): Procedure: Capsulotomy in Direct Anterior Total Hip Arthroplasty
  Interventions: Procedure: Capsulotomy in Direct Anterior Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Capsulectomy in Direct Anterior Total Hip Arthroplasty — Surgical intervention in which the surgeon will perform anterior capsulectomy during total hip arthroplasty.
  Arms: Capsulectomy
Procedure: Capsulotomy in Direct Anterior Total Hip Arthroplasty — Surgical intervention in which the surgeon will perform anterior capsulotomy during total hip arthroplasty. Surgeon will repair the joint capsule.
  Arms: Capsulotomy

SUMMARY:
The purpose of our study is to evaluate the differences in functional activities and proprioception after surgery in subjects who underwent hip prosthesis implant with capsulotomy or capsulectomy.

DETAILED DESCRIPTION:
Concerning hip arthroplasty surgery, in patients affected by coxarthrosis, there are two different techniques: one is capsulectomy and the second one is capsulotomy with repairing the capsule at the end of the procedure. Both preserving and excising the capsule are accepted methods and the choice whether repairing the capsule or not is up to the surgeon, since studies have not yet demonstrated the superiority of one of the two techniques. Articular capsule has a physiological role in joint stability and proprioception. The presence of proprioceptive nerve endings in hip joint capsule has been observed both in healthy patients and in those affected by coxarthrosis.

If capsulectomy is performed during primary hip arthroplasty, the pseudocapsule that is formed in place of the native capsule will not have any active neurophysiological role in the hip.

For this reason, investigators compare the two surgical techniques with the purpose of highlighting, if existing, the superiority of one technique on the other in terms of better functional recovery and proprioceptive sensibility.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral primary hip prosthesis utilizing direct anterior approach
* Age ≥ 18
* Signature of the informed consent

Exclusion Criteria:

* Documented peripheral neuropathies
* Documented central nervous system diseases that may compromise the balance and/or proprioception
* Presence of other joint prosthesis in the lower limbs
* Revision hip arthroplasty
* Symptomatic osteoarthritis of other joints in the lower limbs (including the controlateral hip) or the spine
* BMI > 35
* Systemic diseases or clinical conditions that could interfere with the clinical study
* Neuromuscular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)

SECONDARY OUTCOMES:
Change in Six minutes walk test distance | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
Change in Six minutes walk test distance | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
Change in 30 seconds chair stand test | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
Change in 30 seconds chair stand test | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
Hip Proprioception Evaluation Flexion - Measure of the absolute difference between the actual and the subject-replicated target positions. | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
  Measures of hip flexion repositioning error (active and passive repositioning)
Hip Proprioception Evaluation Abduction - Measure of the absolute difference between the actual and the subject-replicated target positions. | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
  Measures of hip abduction repositioning error (active and passive repositioning)
Hip Proprioception Evaluation External Rotation- Measure of the absolute difference between the actual and the subject-replicated target positions. | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
  Measures of hip external rotation repositioning error (active and passive repositioning)
Hip Proprioception Evaluation Flexion- Measure of the absolute difference between the actual and the subject-replicated target positions. | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
  Measures of hip flexion repositioning error (active and passive repositioning)
Hip Proprioception Evaluation Abduction - Measure of the absolute difference between the actual and the subject-replicated target positions. | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
  Measures of hip abduction repositioning error (active and passive repositioning)
Hip Proprioception Evaluation External Rotation- Measure of the absolute difference between the actual and the subject-replicated target positions. | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
  Measures of hip external rotation repositioning error (active and passive repositioning)
Active hip Range Of Motion Flexion- degree | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
  Measures of hip flexion maximal active Range of Motion
Active hip Range Of Motion Abduction- degree | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
  Measures of hip abduction maximal active Range of Motion
Active hip Range Of Motion External Rotation- degree | Before surgery (T0), 50 days (plus or minus 3 days) after surgery (T1)
  Measures of hip external rotation maximal active Range of Motion
Active hip Range Of Motion Flexion- degree | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
  Measures of hip flexion maximal active Range of Motion
Active hip Range Of Motion Abduction- degree | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
  Measures of hip abduction maximal active Range of Motion
Active hip Range Of Motion External Rotation- degree | Before surgery (T0), 90 days (plus or minus 3 days) after surgery (T2)
  Measures of hip external rotation maximal active Range of Motion
Surgical time- minutes | The day of the surgical procedure
  This will be measured from the time of incision to the time the dressing is applied
Percent hemoglobin drop | Up to 2 weeks after surgery (during inpatient stay)
  Percent hemoglobin drop will be measured by comparing the preoperative hemoglobin to the inpatient nadir hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ometti, MD, Study Director — IRCCS San Raffaele
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hewitt JD, Glisson RR, Guilak F, Vail TP. The mechanical properties of the human hip capsule ligaments. J Arthroplasty. 2002 Jan;17(1):82-9. doi: 10.1054/arth.2002.27674. PMID 11805930
- [Background] Martin HD, Savage A, Braly BA, Palmer IJ, Beall DP, Kelly B. The function of the hip capsular ligaments: a quantitative report. Arthroscopy. 2008 Feb;24(2):188-95. doi: 10.1016/j.arthro.2007.08.024. Epub 2007 Nov 26. PMID 18237703
- [Background] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Background] Moraes MR, Cavalcante ML, Leite JA, Macedo JN, Sampaio ML, Jamacaru VF, Santana MG. The characteristics of the mechanoreceptors of the hip with arthrosis. J Orthop Surg Res. 2011 Nov 16;6:58. doi: 10.1186/1749-799X-6-58. PMID 22087603
- [Background] Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S350-70. doi: 10.1002/acr.20538. No abstract available. PMID 22588756
- [Background] Nilsdotter AK, Lohmander LS, Klassbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC Musculoskelet Disord. 2003 May 30;4:10. doi: 10.1186/1471-2474-4-10. Epub 2003 May 30. PMID 12777182
- [Derived] Ometti M, Brambilla L, Gatti R, Tettamanti A, La Cava T, Pironti P, Fraschini G, Salini V. Capsulectomy vs capsulotomy in total hip arthroplasty. Clinical outcomes and proprioception evaluation: Study protocol for a randomized, controlled, double blinded trial. J Orthop. 2019 Sep 12;16(6):526-533. doi: 10.1016/j.jor.2019.09.020. eCollection 2019 Nov-Dec. PMID 31680746